CLINICAL TRIAL: NCT06003179
Title: Optimizing Lymphodepletion to Improve Outcomes in Patients Receiving Anti Cluster of Differentiation Antigen 19 (Anti-CD19) Chimeric Antigen Receptor T (CAR T) Cell Therapy With Kymriah/tIsagenlecleucel (LOKI)
Brief Title: Optimizing Lymphodepletion to Improve Outcomes in Patients Receiving Cell Therapy With Kymriah
Acronym: LOKI
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: recruitment challenges and sites who initially expressed interest declined.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OZM-123
Record Dates: First submitted 2023-07-10; First posted 2023-08-21 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Intervention Model Description: Patients will be enrolled in two stages: the dose escalation stage to assess the safety and tolerability of a modified LD regimen, and once the maximum tolerated dose (MTD) is determined, a cohort expansion phase to further characterize the toxicity and efficacy profile and determine the recommended phase 2 dose (RP2D). The study will enroll approximately 20-40 patients in the dose escalation stage (Part 1), and approximately 20 further patients at cohort expansion (Part 2).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cyclophosphamide and fludarabine, standard dose (Active Comparator): Fludarabine 25mg/m2 Cyclophosphamide 250mg/m2 Days -4, -3, -2
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine
- Cyclophosphamide and fludarabine, standard dose with radiation (Experimental): Fludarabine 25mg/m2 Cyclophosphamide 250mg/m2 Days -6, -5, -4 2 Gy in 2 Fractions Days -3, -2
  Interventions: Radiation: TLI; Drug: Fludarabine
- Cyclophosphamide (intermediate dose) and fludarabine (Experimental): Fludarabine 25mg/m2 Cyclophosphamide 500mg/m2 Days -4, -3, -2
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine
- Cyclophosphamide (intermediate dose) and fludarabine with radiation (Experimental): Fludarabine 25mg/m2 Cyclophosphamide 500mg/m2 Days -6, -5, -4 2 Gy in 2 Fractions Days -3, -2
  Interventions: Drug: Cyclophosphamide; Radiation: TLI; Drug: Fludarabine
- Cyclophosphamide (high dose) and fludarabine (Experimental): Fludarabine 25mg/m2 Cyclophosphamide 750mg/m2 Days -4, -3, -2
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine
- Cyclophosphamide (high dose) and fludarabine with radiation (Experimental): Fludarabine 25mg/m2 Cyclophosphamide 750mg/m2 Days -6, -5, -4 2 Gy in 2 Fractions Days -3, -2
  Interventions: Drug: Cyclophosphamide; Radiation: TLI; Drug: Fludarabine

INTERVENTIONS:
Drug: Cyclophosphamide — Conditioning chemo at different doses
  Other Names: Cytoxan, neosar
  Arms: Cyclophosphamide (high dose) and fludarabine; Cyclophosphamide (high dose) and fludarabine with radiation; Cyclophosphamide (intermediate dose) and fludarabine; Cyclophosphamide (intermediate dose) and fludarabine with radiation; Cyclophosphamide and fludarabine, standard dose
Radiation: TLI — radiation given with conditioning chemo
  Arms: Cyclophosphamide (high dose) and fludarabine with radiation; Cyclophosphamide (intermediate dose) and fludarabine with radiation; Cyclophosphamide and fludarabine, standard dose with radiation
Drug: Fludarabine — Fludarabine given as part of standard treatment

SUMMARY:
This is a Phase 1b study of participants with Diffuse Large B Cell Lymphoma (DLBCL). The purpose of this study is to identify an optimized lymphodepletion (LD) regimen by evaluating standard and intermediate doses of Fludarabine (Flu) / Cyclophosphamide (Cy) with or without a fixed dose of total lymphoid irradiation (TLI) in the setting of standard of care chimeric antigen receptor T (CAR T) cell therapy.

DETAILED DESCRIPTION:
Patients will be enrolled in two stages: the dose escalation stage to assess the safety and tolerability of a modified LD regimen, and once the maximum tolerated dose (MTD) is determined, a cohort expansion phase to further characterize the toxicity and efficacy profile and determine the recommended phase 2 dose (RP2D). The study will enroll approximately 20-40 patients in the dose escalation stage (Part 1), and approximately 20 further patients at cohort expansion (Part 2). There will be six dose escalation cohorts, in three study arms. There are two dosing cohorts in each study arm. Patients in Arm 1 will receive the JULIET chemotherapy LD regimen with or without TLI, and in Arms 2 and 3, intermediate doses of Cy with a fixed dose of Flu, with or without TLI, will be given.

The cohorts in Arm 1 will enroll concurrently, and enrollment into Arm 2 will begin after Arm 1 has enrolled all patients and data review by the Trial Steering Committee (TSC). Similarly, enrollment into Arm 3 will only commence once Arm 2 has accrued and relevant safety data has been reviewed.

For accrual into Cohort 2, Arm 1, there will be a 15-day staggered enrollment for the first 2 patients. Staggered enrollment with another 15-day delay may be considered for enrollment into relevant cohorts in Arms 2 and 3, after review by the TSC.

Following completion of accrual to Arm 1, a 30 day dose limiting toxicity (DLT) window will be observed, prior to review by the TSC and commencement of patient enrollment into Arm 2. The same procedure and DLT window will be followed prior to patient enrollment into Arm 3.

One DLT window will be observed during this study: 30 days post infusion of tisagenlecleucel.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of informed consent
2. Life expectancy ≥ 12 weeks
3. Biopsy-proven and histologically confirmed relapse/refractory (R/R) large B cell lymphoma, including Primary mediastinal B-cell lymphoma (PMBCL), R/R DLBCL and transformation from Follicular lymphoma (FL).
4. Radiographically documented measurable disease as per Lugano response criteria (i.e. longest transverse diameter of a lesion (LDi) > 1.5 cm that is [18F] fluorodeoxyglucose (FDG) avid).
5. At least 2 weeks or 5 half-lives, whichever is shorter, must have elapsed since any prior systemic cancer therapy at the time the subject provides consent
6. Eligible for standard of care CAR T cell therapy, specifically, relapsed or refractory large B cell lymphoma after two or more lines of systemic therapy, and subjects must have received adequate first-line therapy including at a minimum:
7. Patient is sufficiently stable to facilitate planned CAR T-cell therapy (e.g. not rapidly progressing on temporizing therapy, no significant compromise of vital organ functions (intubation, dialysis, requiring Intensive care unit (ICU)/vasopressor support)) and has good performance status
8. Patient does not have active central nervous system (CNS) disease
9. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 at enrollment
10. Patient has not received prior adoptive T-cell immunotherapy
11. Patient is not human immunodeficiency virus (HIV) positive
12. Patient did not receive prior allogeneic stem cell transplant
13. Adequate bone marrow, renal, hepatic, pulmonary and cardiac function
14. Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential)
15. Sexually active males who accept to use a condom during intercourse during treatment and for 12 months after treatment as they should not father a child in this period. A condom is required to be used also by vasectomized men (as well as during intercourse with a male partner) in order to prevent delivery of the drug via seminal fluid
16. Must have an apheresis product of non-mobilized cells accepted for manufacturing.

Exclusion Criteria:

1. Persisting disease bulk (defined as ≥10 cm) on restaging imaging following bridging therapy.
2. History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) unless disease free for at least 3 years
3. History of Richter's transformation of chronic lymphocytic leukemia (CLL)
4. History of allogeneic stem cell transplant
5. Received < 2 lines of therapy for large B cell lymphoma
6. Prior CD19 targeted therapy
7. Subject has received or undergone the protocol defined treatments/therapies
8. Prior chimeric antigen receptor therapy or other genetically modified T-cell therapy
9. Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring intravenous (IV) antimicrobials for management. Simple urinary tract infection (UTI) and uncomplicated bacterial pharyngitis are permitted if responding to active treatment.
10. Known history of infection with human immunodeficiency virus (HIV) or hepatitis B (HBsAg positive) or hepatitis C virus (anti-HCV positive). If there is a positive history of treated hepatitis B or hepatitis C, the viral load must be undetectable per quantitative polymerase chain reaction (PCR) and/or nucleic acid testing.
11. Active tuberculosis
12. Subjects with detectable cerebrospinal fluid malignant cells or known CNS involvement; a history of prior treated CNS lymphoma which is not active at the time of relapse is permitted
13. History or presence of significant non-malignant CNS disorder such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement
14. Subjects with cardiac atrial or cardiac ventricular lymphoma involvement
15. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, New York Heart Association Class II or greater congestive heart failure, or other clinically significant cardiac disease within 12 months of enrollment
16. Requirement for urgent therapy due to tumor mass effects such as bowel obstruction or blood vessel compression
17. History of autoimmune disease, requiring systemic immunosuppression and/or systemic disease modifying agents within the last 2 years.
18. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis per chest computed tomography (CT) scan at screening. History of radiation pneumonitis in the radiation field (fibrosis) is allowed.
19. History of symptomatic deep vein thrombosis or pulmonary embolism within 6 months of enrollment
20. Any medical condition likely to interfere with assessment of safety or efficacy of study treatment
21. History of severe immediate hypersensitivity reaction to tocilizumab or any of the agents used in this study
22. Treatment with a live, attenuated vaccine within 6 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during the course of the study
23. Women of childbearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of chemotherapy on the fetus or infant.
24. Subjects of either sex who are not willing to practice birth control from the time of consent and at least 6 months after tisagenlecleucel infusion
25. In the investigators judgment, the subject is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and dose limiting toxicity (DLT) for chemo plus radiation as lymphodepletion | baseline through end of study completion, approximately 2 years
  (LD) regimen (Fludarabine (Flu)/Cyclophosphamide (Cy) + total lymphoid irradiation (TLI ) in patients receiving standard of care CAR T cell therapy for relapsed/refractory diffuse large B cell lymphoma (R/R DLBCL) by establishing the maximum tolerated doses (MTD) of standard (JULIET) dose Flu/Cy + TLI, and of intermediate dose iCy/Flu +/- TLI and the dose limiting toxicities (DLT) of standard dose Flu/Cy + TLI, and of intermediate dose iCy/Flu +/- TLI

SECONDARY OUTCOMES:
overall response rate (ORR) at 12 months of chemo rads | baseline to 12 months post CAR-T
  To assess the ORR at 12 months of a combination chemo-radiation LD regimen (standard dose Flu/Cy + TLI) in patients receiving CAR T cell therapy for R/R DLBCL.
complete response (CR) rate at 12 months of chemo rads | baseline to 12 months post CAR-T
  To assess the CR rate of a combination chemo-radiation LD regimen (standard dose Flu/Cy + TLI) in patients receiving CAR T cell therapy for R/R DLBCL.
progression free survival (PFS) at 12 months of chemo rads | baseline to 12 months post CAR-T
  To assess the PFS rate at 12 months of a combination chemo-radiation LD regimen (standard dose Flu/Cy + TLI) in patients receiving CAR T cell therapy for R/R DLBCL.
ORR at 12 months of an intermediate dose iCy/Flu +/- TLI LD regimen | baseline to 12 months post CAR-T
  To assess the ORR at 12 months of an intermediate dose iCy/Flu +/- TLI LD regimen in patients receiving CAR T cell therapy for R/R DLBCL
CR rate at 12 months of an intermediate dose iCy/Flu +/- TLI LD regimen | baseline to 12 months post CAR-T
  To assess the CR rate at 12 months of an intermediate dose iCy/Flu +/- TLI LD regimen in patients receiving CAR T cell therapy for R/R DLBCL
PFS at 12 months of an intermediate dose iCy/Flu +/- TLI LD regimen | baseline to 12 months post CAR-T
  To assess the PFS rate at 12 months of an intermediate dose iCy/Flu +/- TLI LD regimen in patients receiving CAR T cell therapy for R/R DLBCL

OTHER OUTCOMES:
Assessments | During lymphodepleting therapy
  To define the appropriate dose to be administered weight in kilograms and height in meters will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: John G Kuruvilla, Principal Investigator — Princess Margaret Cancer Centre - University Health Network
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada